CLINICAL TRIAL: NCT03517592
Title: A Multicenter Phase II Rater-Blinded Randomized Controlled Trial to Compare the Effectiveness of Eye Movement Desensitization Reprocessing Therapy vs. Treatment as Usual in Patients With Substance Use Disorder and History of Psychological Trauma
Brief Title: EMDR Versus Treatment As Usual in Patients With Substance Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/7615/I
Record Dates: First submitted 2018-04-04; First posted 2018-05-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-03

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR Therapy (Experimental): EMDR: 20 individual sessions 60 minutes each for 6 months
  Interventions: Other: EMDR
- Treatment as Usual (Other): The TAU condition includes follow-up visits with the psychiatry, psychology and with the nursing service. Visits with the psychiatrist consist to evaluate clinical status and readjust the pharmacological treatment if necessary while visits with the psychologist consist to assess and detect risk situations and to prevent relapses using a cognitive behavioral approach. Finally, the nursing service will provide health and care habits and will carry out the abstinence controls.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: EMDR — The EMDR SUD Protocol consists of a detailed interview with respect to traumatic events, the treatment of those with the EMDR standard protocol and a further specific protocol for SUD that is focused on the concept of addiction memory.
  Arms: EMDR Therapy
Other: Treatment as Usual — The TAU condition includes follow-up visits with the psychiatry, psychology and with the nursing service. Visits with the psychiatrist consist to evaluate clinical status and readjust the pharmacological treatment if necessary while visits with the psychologist consist to assess and detect risk situations and to prevent relapses using a cognitive behavioral approach. Finally, the nursing service will provide health and care habits and will carry out the abstinence controls.
  Arms: Treatment as Usual

SUMMARY:
The main objective of this project is to test whether EMDR therapy is effective in reducing substance use and improving clinical and trauma-related symptoms in SUD patients with a history of psychological trauma.

DETAILED DESCRIPTION:
Background:

Substance use disorders (SUD) represent an important social and public health problem due to their negative consequences in terms of delinquency, family disintegration, academic and occupational disengagement, mental illness, transmission of infectious diseases, intoxication and mortality rates. As with other mental disorders, the evolution of this disorder depends on many biological and sociodemographic variables, such as the age of onset of consumption, access to drugs, one's living environment, race, and the presence of stressors. Of all these variables, adverse events are being increasingly investigated, due to the strong negative impact they have on the onset, course and prognosis of psychiatric disorders, especially when psychological trauma is present. Traumatic events, especially in childhood or adolescence, are considered to be a robust risk factor for developing post-traumatic stress disorder (PTSD), with or without further comorbid severe mental disorders such as depression, bipolar disorder, psychosis or SUD. A recent meta-analysis published in the Lancet found multiple adverse childhood events to be a significant risk factor for problematic alcohol and substance use, highlighting the impact of adverse childhood events even when not associated with a diagnosis of PTSD. Although there is currently no available data about the prevalence of traumatic events in SUD patients population, it is estimated that is likely high presumed to be high. The results of different studies estimate that the prevalence of PTSD in inpatients with SUD to ranges from 25% -51%, which is two to four times higher than the prevalence range found in the general population (1.3% -12.3%). In addition, evidence suggests that PTSD and traumatic events are correlated with addiction severity, with a worse disease prognosis, with a greater number of hospitalizations, with a poorer response to treatment, with shorter periods of abstinence and with greater craving. Thus, an integral model with an individualized treatment plan is indicated in SUD, including psychological trauma as a specific objective to address.

A possible candidate for this is Eye Movement Desensitization and Reprocessing (EMDR) therapy, which is considered to be a first line treatment for PTSD, being recommended by different international bodies, such as the American Psychiatric Association (APA) and World Health Organization (WHO). EMDR is a psychotherapeutic approach designed to alleviate the distress associated with traumatic memories, facilitating the access to and processing of traumatic memories and other adverse life experiences and bringing these to an adaptive resolution using standardized protocols and elements of cognitive behavioral, interpersonal, and body-centered therapies in conjunction with bilateral stimulation (e.g. horizontal eye movements from side to side). In recent years, the use of EMDR has increased exponentially in clinical practice due its effectiveness and safety and that has resulted in investigations in additional populations beyond PTSD, such as in those with depression, anxiety, chronic pain, bipolar disorder, or psychosis. Of note, three small randomized controlled trials (RCT) of EMDR versus Treatment As Usual (TAU) have also been performed in patients with SUD. The results suggest that EMDR, compared to the control group, significantly improved craving, depression, anxiety, self-esteem and dissociative symptoms, but samples were small. A large scale RCT is currently underway, which aims to determine the efficacy of EMDR in reducing PTSD symptoms in an inpatient sample with comorbid PTSD or subthreshold PTSD and SUD. In view of the above, we consider that a further large RCT of EMDR in the treatment of psychological trauma in outpatients with SUD, including psychological trauma related to adverse events not covered by DSM-V diagnostic criteria, is crucial and clinically necessary due to the negative impact it has on the course and prognosis of these illnesses, and in order to confirm or reject prior first positive evidence. Our study is also important in including patients with dual pathology and measuring impact on psychopathological symptoms, which will help facilitate the application of EMDR in a real world setting if it is shown to be efficacious.

Design:

This is a single-blind RCT with two parallel branches, EMDR and TAU, in patients diagnosed with SUD who have suffered from comorbid psychological trauma. The patients will be matched by center, age, sex and diagnosis. One group will consist of TAU + 20 individual EMDR sessions, 60 minutes each, during 6 months, the other group will receive TAU only. Patients will be evaluated at baseline, at 3 months, post-treatment at 6 months and at 12 months as follow-up.

Clinical and diagnostic variables:

1. Clinical diagnosis of the participants will employ DSM-V criteria for SUD based on clinical interview (Psychiatric Research Interview for Substance and Mental Disorders; PRISM). The investigators also will use the Mini-International Neuropsychiatric Interview for the detection of the most frequent comorbid psychiatric diagnoses in substance abusers.
2. Clinical Severity of the participants will be assessed by different instruments:

   1. Hamilton Depression Rating Scale: It has been designed to assess the severity and changes of depressive symptoms.
   2. Young Mania Rating Scale:It is a hetero-administered scale composed of 11 items aimed at quantifying the severity of manic and hypo manic episodes.
   3. Brief Psychiatric Rating Scale: It is a hetero-administered scale composed of 18 items measuring psychopathological changes. It includes anxious, affective and psychotic symptoms with each symptom rated on a severity scale of 1-7.

The consumption of SUD is quantified using the following tools:

1. Timeline Followback Questionnaire.
2. Severity of Dependence Scale.
3. Visual Analog Scale.

Trauma symptoms and overall functioning will be evaluated by the following instruments:

1. Childhood Trauma Questionnaire.
2. The Holmes-Rahe Life Stress Inventory.
3. Impact of Event Scale - Revised.
4. Subjective Unit of Discomfort.
5. Dissociative Experiences Scale.
6. Functioning Assessment Short Test: This is a brief instrument to evaluate performance in six different areas of functioning, such as autonomy, occupational functioning, cognitive functioning, finances, relationships and leisure.

The investigators have included a Spanish validated version of all these instruments.

Statistical analysis:

1. Computation of sample size: The study aims to assess the efficacy of EMDR therapy compared with TAU for patients with SUD focused on reduction of substance use, reduction of symptoms associated with craving, associated symptoms of anxiety and depression and functioning. The sample size has been calculated based on a comparison of a normal variable (pre-post reduction) between two independent groups (treated and untreated) using the statistical package R (http: //www.r-project.org/), using an alpha = 0.005 instead of 0.05 to allow correction for multiple comparisons. The number of patients required to detect major effects (d = 0.8) with a statistical power of 80% and alpha = 0.005 is n = 60 per intervention group (two groups, n total = 120). Assuming a loss percentage of approximately 10-15% of the patients in the study, it would be necessary to recruit approximately 132 patients, 66 for each intervention branch.
2. Analysis of the main variables: The distribution of socio-demographic and clinical characteristics between groups in the baseline state will be analyzed by means of descriptive statistics. The continuous variables with a normal distribution will be analyzed with the Analysis of Multivariate Variation (ANOVA). The change in clinical and functional variables with regard to baseline evaluation at strategic points of the intervention will be analyzed using linear models of mixed effects and repeated measures, including fixed factors of time, treatment conditions and their interaction, and the random center factor. The differences between groups, for the categorical variables and main clinics, will be analyzed by adding covariates to the models. Those covariates that are statistically significant may be added in the same model to determine which covariates are best predictors of the response. The index of the size of the effect (index g of Hedges or r of Pearson) of each of the analysis carried out will be estimated. It will be corrected for multiple comparisons. The statistical software used for the analysis will be the latest available version of the SPSS (version 23).
3. Analysis of clinical efficacy: For the main statistical analysis, the population will be used for intent to treat (ITT). The "Last Observation Carried Forward" (LOCF) method will be used as a measure of minimization of lost ones.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* outpatients
* presence of one or more traumatic events, which causes currently trauma associated symptoms (Scale of the impact of the event-reviewed, IES-R> 0) and subjective Disability Unit (SUD)>5)

Exclusion Criteria:

* presence of organic brain diseases
* presence of suicidal ideas
* having received a trauma focused therapy in the last 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in severity of consumption | Changes from baseline to visits at 3, 6 and 12 months.
  To measure changes in the Severity of Dependence Scale. 4-point Likert scale (0 - 3). The higher score indicate greater dependence.
Reduction in level of consumption | Changes from baseline to visits at 3, 6 and 12 months.
  To measure changes in the Visual Analog Scale. It ranges from 0 to 10: the higher the score, the greater the craving severity.
Reduction in the number of relapses | Change of relapses from baseline to visits at 3, 6 and 12 months.
  To measure relapses with the Timeline Followback Questionnaire. It is a retrospective calendar-based measure of daily substance use.
Reduction of (hypo) manic symptoms associated with a comorbid psychiatric disorder | Changes from baseline to visits at 6 and 12 months.
  To measure changes in the Young Mania Rating Scale. It ranges from 0 to 130: the higher the score, the worse the manic symptoms.
Reduction of general psychopathological symptoms associated with psychiatric comorbidity | Change from baseline to visits at 6 and 12 months.
  To measure changes in the Brief Psychiatric Rating Scale. It ranges from 18 to 126: the higher the score, the worse the general psychopathology symptoms.
Reduction in depressive symptoms associated with a comorbid psychiatric disorder | Changes from baseline to visits at 6 and 12 months.
  To measure changes in the Hamilton Depression Rating Scale. Total scores range from 0 to 52: the higher the score, the worse the depressive symptoms.

SECONDARY OUTCOMES:
Improvement of global functioning | Changes from baseline to visits at 6 and 12 months.
  To measure changes with the Functioning Assessment Short Test. The global score ranges from 0 to 72. The higher the score, the poorer the functional status.
Detection of Childhood life traumatic events | Childhood. It is administered only during the baseline visit.
  To assess life events with the Childhood Trauma Questionnaire. A 5-point Likert scale is used, ranging from "Never True" to "Very Often True".
Detection of traumatic events in the last year | The last year. It is administered only during the baseline visit.
  To assess events with The Holmes-Rahe Life Stress Inventory. Scores below 150 reflect low levels of stress, scores between 150 and 299 represent a 50% risk of a stress-related illness in the near future and scores above 300 represent an 80% risk.
Making a PTSD diagnosis | Changes from baseline to visits at 6 and 12 months.
  To diagnose PTSD with the Global Assessment of Posttraumatic Stress Questionnaire. Higher scores indicate more severity in trauma-related symptoms.
Assessment of the severity of trauma-related symptoms. | The previous 7 days. Changes from baseline to visits at 6 and 12 months.
  To measure severity and changes in trauma-related symptoms with the Impact of Event Scale - Revised. Items are rated on a 5-point Likert scale ranging from 0 and 4, yielding a total score ranging from 0 to 88.
Detection of dissociative symptoms | Changes from baseline to visits at 6 and 12 months.
  To assess dissociative symptoms with the Dissociative Experiences Scale. An overall mean score ranging from 0 to 100. The higher score, the higher the severity of the dissociative symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt L Amann, PhD, MD, Principal Investigator — Parc de Salut Mar
Locations (2):
- Spain (2):
  - Germanas Hospitalarias Benito Menni, Sant Boi de Llobregat, Barcelona
  - Parc de Salut Mar, Barcelona

REFERENCES:
- [Background] Driessen M, Schulte S, Luedecke C, Schaefer I, Sutmann F, Ohlmeier M, Kemper U, Koesters G, Chodzinski C, Schneider U, Broese T, Dette C, Havemann-Reinecke U; TRAUMAB-Study Group. Trauma and PTSD in patients with alcohol, drug, or dual dependence: a multi-center study. Alcohol Clin Exp Res. 2008 Mar;32(3):481-8. doi: 10.1111/j.1530-0277.2007.00591.x. Epub 2008 Jan 22. PMID 18215214
- [Background] Mauritz MW, Goossens PJ, Draijer N, van Achterberg T. Prevalence of interpersonal trauma exposure and trauma-related disorders in severe mental illness. Eur J Psychotraumatol. 2013;4. doi: 10.3402/ejpt.v4i0.19985. Epub 2013 Apr 8. PMID 23577228
- [Background] Gradus JL. Prevalence and prognosis of stress disorders: a review of the epidemiologic literature. Clin Epidemiol. 2017 May 3;9:251-260. doi: 10.2147/CLEP.S106250. eCollection 2017. PMID 28496365
- [Background] Kok T, de Haan H, van der Meer M, Najavits L, de Jong C. Assessing traumatic experiences in screening for PTSD in substance use disorder patients: what is the gain in addition to PTSD symptoms? Psychiatry Res. 2015 Mar 30;226(1):328-32. doi: 10.1016/j.psychres.2015.01.014. Epub 2015 Jan 28. PMID 25687377
- [Background] Novo P, Landin-Romero R, Radua J, Vicens V, Fernandez I, Garcia F, Pomarol-Clotet E, McKenna PJ, Shapiro F, Amann BL. Eye movement desensitization and reprocessing therapy in subsyndromal bipolar patients with a history of traumatic events: a randomized, controlled pilot-study. Psychiatry Res. 2014 Sep 30;219(1):122-8. doi: 10.1016/j.psychres.2014.05.012. Epub 2014 May 15. PMID 24880581
- [Background] Shapiro F. The role of eye movement desensitization and reprocessing (EMDR) therapy in medicine: addressing the psychological and physical symptoms stemming from adverse life experiences. Perm J. 2014 Winter;18(1):71-7. doi: 10.7812/TPP/13-098. PMID 24626074
- [Background] Novo Navarro P, Landin-Romero R, Guardiola-Wanden-Berghe R, Moreno-Alcazar A, Valiente-Gomez A, Lupo W, Garcia F, Fernandez I, Perez V, Amann BL. 25 years of Eye Movement Desensitization and Reprocessing (EMDR): The EMDR therapy protocol, hypotheses of its mechanism of action and a systematic review of its efficacy in the treatment of post-traumatic stress disorder. Rev Psiquiatr Salud Ment (Engl Ed). 2018 Apr-Jun;11(2):101-114. doi: 10.1016/j.rpsm.2015.12.002. Epub 2016 Feb 11. English, Spanish. PMID 26877093
- [Background] Hase M, Balmaceda UM, Hase A, Lehnung M, Tumani V, Huchzermeier C, Hofmann A. Eye movement desensitization and reprocessing (EMDR) therapy in the treatment of depression: a matched pairs study in an inpatient setting. Brain Behav. 2015 Jun;5(6):e00342. doi: 10.1002/brb3.342. Epub 2015 Apr 30. PMID 26085967
- [Background] Behnammoghadam M, Alamdari AK, Behnammoghadam A, Darban F. Effect of Eye Movement Desensitization and Reprocessing (EMDR) on Depression in Patients With Myocardial Infarction (MI). Glob J Health Sci. 2015 Apr 19;7(6):258-62. doi: 10.5539/gjhs.v7n6p258. PMID 26153191
- [Background] Feske U, Goldstein AJ. Eye movement desensitization and reprocessing treatment for panic disorder: a controlled outcome and partial dismantling study. J Consult Clin Psychol. 1997 Dec;65(6):1026-35. doi: 10.1037//0022-006x.65.6.1026. PMID 9420364
- [Background] Doering S, Ohlmeier MC, de Jongh A, Hofmann A, Bisping V. Efficacy of a trauma-focused treatment approach for dental phobia: a randomized clinical trial. Eur J Oral Sci. 2013 Dec;121(6):584-93. doi: 10.1111/eos.12090. Epub 2013 Sep 23. PMID 24206075
- [Background] Nazari H, Momeni N, Jariani M, Tarrahi MJ. Comparison of eye movement desensitization and reprocessing with citalopram in treatment of obsessive-compulsive disorder. Int J Psychiatry Clin Pract. 2011 Nov;15(4):270-4. doi: 10.3109/13651501.2011.590210. Epub 2011 Aug 3. PMID 22122001
- [Background] Gerhardt A, Leisner S, Hartmann M, Janke S, Seidler GH, Eich W, Tesarz J. Eye Movement Desensitization and Reprocessing vs. Treatment-as-Usual for Non-Specific Chronic Back Pain Patients with Psychological Trauma: A Randomized Controlled Pilot Study. Front Psychiatry. 2016 Dec 20;7:201. doi: 10.3389/fpsyt.2016.00201. eCollection 2016. PMID 28066274
- [Background] Perez-Dandieu B, Tapia G. Treating Trauma in Addiction with EMDR: A Pilot Study. J Psychoactive Drugs. 2014 Oct-Dec;46(4):303-9. doi: 10.1080/02791072.2014.921744. PMID 25188700
- [Result] Tirado-Munoz J, Gilchrist G, Fischer G, Taylor A, Moskalewicz J, Giammarchi C, Kochl B, Munro A, Dabrowska K, Shaw A, Di Furia L, Leeb I, Hopf C, Torrens M. Psychiatric comorbidity and intimate partner violence among women who inject drugs in Europe: a cross-sectional study. Arch Womens Ment Health. 2018 Jun;21(3):259-269. doi: 10.1007/s00737-017-0800-3. Epub 2017 Dec 11. PMID 29230558
- [Derived] Valiente-Gomez A, Moreno-Alcazar A, Radua J, Hogg B, Blanco L, Lupo W, Perez V, Robles-Martinez M, Torrens M, Amann BL. A Multicenter Phase II Rater-Blinded Randomized Controlled Trial to Compare the Effectiveness of Eye Movement Desensitization Reprocessing Therapy vs. Treatment as Usual in Patients With Substance Use Disorder and History of Psychological Trauma: A Study Design and Protocol. Front Psychiatry. 2019 Mar 15;10:108. doi: 10.3389/fpsyt.2019.00108. eCollection 2019. PMID 30930801